CLINICAL TRIAL: NCT05507723
Title: Effect of Tight Urate Control in Gouty Arthritis Compared to Usual Care (TICOGA), a Randomised Clinical Trial
Brief Title: Tight Control of Gouty Arthritis Compared to Usual Care
Acronym: TICOGA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: AC22077
Record Dates: First submitted 2022-07-22; First posted 2022-08-19 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Gout
Keywords: treat-to-target; gout
MeSH Terms: conditions — Gout

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treat-to-target (Experimental): All participants will have the GoutSMART application installed on their phones, and be offered a management plan including the use of flare prophylaxis and maximum advised dose of allopurinol based on renal function. All Participants in the treat-to-target group will be provided with a BeneCheck hand-held device and taught to perform urate finger prick self-testing. Participants will be prompted to submit urate readings by the GoutSMART app and if urate levels remain above target their allopurinol will be increased incrementally up to the pre-specified maximum dose of allopurinol.
  Interventions: Other: Treat-to-target
- Usual care (Active Comparator): All participants will have the GoutSMART application installed on their phones, and be offered a management plan including the use of flare prophylaxis and maximum advised dose of allopurinol based on renal function to achieve urate target. Participants in the usual care arm of the study will have their treatment reviewed and escalated by their GPs in line with usual practice.
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Treat-to-target — Treatment to achieve urate target using supported self-management approach
  Arms: Treat-to-target
Other: Usual Care — Treatment escalation by GP based on usual clinical practice
  Arms: Usual care

SUMMARY:
Gout is caused by a reaction to urate crystals that results in attacks of severe joint pain. Medicines that lower urate levels can prevent gout flares, however it takes time for this benefit to be felt, and paradoxically starting treatment with large doses of urate lowering treatment risks provoking attacks of gout. Medical guidelines disagree on the best way to overcome these challenges with many recommending medicine dose adjustment based on regular urate testing but a general practice guideline suggesting more simply increasing the medicine dose in those patients that continue to suffer flares. In reality most patients are not treated at all, and many of those that are treated never receive an effective dose of treatment. We have developed a supported self-management approach to gout in which patients monitor their own urate levels using a finger prick test, and then receive advice on adjusting their treatment dose to achieve target urate levels through a smartphone app (Gout SMART). A trial of this approach has shown that it results in much better control of urate levels after 6 months than usual care, and suggests that it also leads to fewer flares. We would now like to confirm that this approach is effective in reducing flares of gout over 2 years by randomising patients to either treatment-to-target urate using our self-monitoring approach, or to usual care.

DETAILED DESCRIPTION:
A total of approximately 120 participants will be recruited. We anticipate that most participants will be identified following referral to rheumatology outpatient or on-call services in National Health Service (NHS) Lothian, or through NHS Lothian's gout liaison service. Additional patients may indicate their willingness to participate directly in response to study advertisements.

Based on baseline renal function and flare frequency, an individual treatment plan will be drawn up for all participants which will set a ceiling on the maximum dose of allopurinol to be used within the trial and determine the need for flare prophylaxis with colchicine. Participants will be randomized to the intervention group in a 1:1 ratio, with stratification by the need for use of flare prophylaxis.

All participants will have a smart phone application (GoutSMART) uploaded to their smart phones. Usual care participants will have a limited version of the GoutSMART application installed which includes background information about gout and provides a means for participants to maintain diaries of gout flares. Subjects in the usual care arm of the study will have treatment escalation decisions made by their GPs. Subjects in the treat-to-target arm will be taught to self-test serum urate using a BeneCheck Plus hand held device and provided with test strips. A full version of the GoutSMART application will be installed with the features mentioned above but also the facility to record a urate diary. Participants will be prompted to check their serum urate and enter the results into the GoutSMART application. Participants reporting a urate level >0.3mmol/l will be advised to increase the dose of allopurinol incrementally as specified in their treatment plan. No change will be advised in those whose urate levels are already at target. If the patient needs to increase allopurinol there will be an automatic reminder after two weeks prompting the patients to submit updated self-test results which will be handled in the same way as described above. Conversely for participants achieving target levels this will be acknowledged and a request to resubmit readings will be sent on a monthly basis.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent.
* Age ≥18 years.
* Patient has sustained at least one flare of gout in the previous 12 months.
* Confirmed clinical diagnosis of gout as per ACR/EULAR criteria
* Serum urate >0.36mm/L.
* Patient has a smart phone and is able to install GoutSMART application.

Exclusion Criteria:

* Subject unable to provide consent
* Patient on maximum urate lowering therapy or where therapy cannot be escalated further due to intolerance/adverse reaction to either allopurinol or febuxostat.
* End stage renal failure/transplant
* Current prescription of medication known to interact with xanthine oxidase inhibitors such as azathioprine or mercapto-purine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-06-12 (Actual); Primary Completion 2028-05-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants flare free in 2nd year of trial | 2nd year of trial
  Proportion of participants flare free in 2nd year of trial

SECONDARY OUTCOMES:
Number of flares of gout | 2 years
  Number of flares of gout in year 1, year 2 and over whole course of trial
Urate targets of ≤0.3mmol/L or ≤0.36mmol/L | 2 years
  Proportion of participants achieving urate levels of ≤0.3mmol/L or ≤0.36mmol/L at 52 and 104wks
Presence of tophi | 2 years
  Proportion of participants with tophi at week 52 and 104
Societal cost | 2 years
  Number of days lost at work and number of medical appointments or hospital admissions due to gout
Time to remission | 2 years
  Time to last flare of gout and time to resolution of tophi
User engagement | 2 years
  User engagement with smartphone app (number of reminders needed for each submission)
Medication prescriptions | 2 years
  Medication compliance assessed by community prescriptions issued
Quality of life using SF-36 questionnaire | 2 years
  Self-reported quality of life at week 52 and week 104 using SF 36 questionnaire. Global health score (0 to 100 score with 100 representing best possible health)
Activity limitation | 2 years
  Functional impact assessed with HAQ-DI questionnaire at week 52 and 104
Medication compliance | 2 years
  Medication compliance assessed by patient self-report at week 52 and 104
Cost-effectiveness | 2 years
  Cost per flare avoided
Cost-Utility | 2 years
  Cost per quality adjusted life year gained
Patient attitudes and understanding | 2 years
  Exploration of patient attitudes and understanding through qualitative interview

CONTACTS AND LOCATIONS:
Overall Officials: Philip L Riches, FRCP, PhD, Principal Investigator — NHS Lothian
Locations (1):
- NHS Lothian, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie results of specified outcomes will be shared after deidentification.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Deidentified information will be made available immediately following publication of trial results and be kept available for 5 years.
Access Criteria: Researchers who provide a methodologically sound proposal.
URL: https://www.ed.ac.uk/centre-genomic-medicine/research-groups/philip-riches/gout-smart

REFERENCES:
- [Background] Riches PL, Alexander D, Hauser B, Kuske B, Krause A. Evaluation of supported self-management in gout (GoutSMART): a randomised controlled feasibility trial. Lancet Rheumatol. 2022 May;4(5):e320-e328. doi: 10.1016/S2665-9913(22)00062-5. Epub 2022 Mar 24. PMID 38294032
- See also: University of Edinburgh trial website — https://www.ed.ac.uk/centre-genomic-medicine/research-groups/philip-riches/gout-smart